CLINICAL TRIAL: NCT01264406
Title: Examination of Mechanisms (E-MECHANIC) of Exercise-induced Weight Compensation
Brief Title: The Comparison of Energy in Take and Body Weight EXERCISE
Acronym: E-MECHANIC
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Corby K. Martin, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 10008
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Results first posted 2024-12-10 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Exercise; Energy; Body Weight
MeSH Terms: conditions — Motor Activity; Body Weight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Exercise Group (20 KKW): Exercise group will obtain 20 KKW, perform in 4-5 sessions per week for approximately 50-70 minutes per session.
- Exercise Group (8 KKW): One exercise group will obtain 8KKW (kcal/kg/week) over 3-4 sessions per wee, which will result in each session lasting approximately 30 minutes
- Control group: This group will be instructed to maintain their baseline level of exercise.

SUMMARY:
This study will compare the effect of two doses of exercise on energy intake and body weight. The comparison will be between three groups; two exercise groups and a control group. The exercise groups will not be provided with a dietary intervention and the study design also includes a non-exercise control group. E-Mechanic trial can make important contributions to understanding of the role of exercise dose in weight management. While it is accepted that regular exercise plays an important role in general health, the exact role of exercise in prevention of weight gain, weight loss and prevention of weight regain remains poorly understood despite exercise being widely prescribed for these purposes. The idea that current weight management exercise recommendations may produce increased energy intake (or other forms on compensation) resulting in disappointing weight loss is an important public health issue. The finding of this study could help shape future exercise and weight loss recommendations and treatment plans.

DETAILED DESCRIPTION:
The purpose of the E-MECHANIC Trial is to test the effect of two doses of exercise on energy intake, body weight, body composition, activity levels, and metabolic rate. The exercise doses will reflect current recommendations for: 1) general health (8 KKW), and 2) weight loss (20 KKW). A non-exercise control group will also be recruited. The primary outcome variables are: 1) energy intake, and 2) the discrepancy between expected weight loss and observed weight loss. Energy intake will be measured using doubly labeled water and laboratory-based food intake tests. Secondary outcome variables include resting metabolic rate, activity levels (excluding structured exercise), and body composition. Following a comprehensive baseline assessment, participants will be randomly assigned to the 8 KKW, 20 KKW, or control group in a 1:1:1 ratio. Additional assessments will be conducted at week 4, with another comprehensive assessment at week 24. The week 4 assessment is important to determine if endpoints change in the short-term, but not long-term.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 - 65 years old, inclusive

  * Not exercising > 20 minutes on > 3 days/wk and taking < 8000 steps/d over one week measured with step counters.
  * BMI > 25 kg/m2 and < 40 kg/m2

Exclusion Criteria:

* • Current consumption of more than 14 alcoholic drinks per week

  * Plan to move out of the study area within the next 6 months or plan to be out of the study area for more than 4 weeks in the next 6 months
  * Have another member of household participating in the study
  * Residence too far from Pennington
  * A past history and/or physical examination or laboratory findings of the following medical conditions:

Table 1. Exclusion Criteria

* Cardiovascular disease (CVD) or disorders Potential participants with a history of CVD
* Blood Pressure Potential participants who are on a stable dose of antihypertensive medication, with the exception of beta-blockers, and whose blood pressure is controlled will be eligible for enrollment.
* Diabetes Potential participants with a previous diagnosis of diabetes (Type 1 or 2) or a fasting plasma glucose >125 mg/dl will be excluded from the study.
* Blood lipids Potential participants whose LDL-C 190 mg/dl or TG levels 300 mg/dl will be referred to their physician.
* Hematologic disorders Participants diagnosed with hematologic disorders, including anemias, bleeding disorders, chronic thrombotic disorders, or hypercoagulable states, will not be allowed into the study.
* Recent blood donation or blood loss Blood donation or blood loss from surgery or trauma during the 6 weeks before the baseline evaluation
* Weight loss-20 or more kilograms in the past year Other exclusions.
* Hospitalization for mental illness within the past 5 years or currently undergoing treatment for severe mental illness. Plans to be out of the city more than 4 weeks over the next 6 months
* Other significant medical conditions Including but not limited to chronic or recurrent respiratory, gastrointestinal, neuromuscular, neurological, or psychiatric conditions. Musculoskeletal problems interfering with exercise.
* Autoimmune or collagen vascular diseases. Immunodeficiency diseases or a positive HIV test. Malignancies in the past 5 years, with the exception of non-melanoma skin cancer therapeutically controlled. Any other medical condition or disease that is life-threatening or that can interfere with or be aggravated by exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population group will be 198 sedentary, overweight and obese(BMI levels > 25 kg/m2 and < 40 kg/m2) individuals. Based on previous studies, we expect to enroll 132 females and 66 males. Participants will be randomly assigned to an 8 kcal/kg/week, 20 kcal/kg/week, or control group. The exercise groups will be closely monitored during exercise sessions for six months in our exercise-training laboratory.
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2010-12; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corby Martin, PhD, Principal Investigator — PBRC; Timothy Church, MD; MPH; PhD, Principal Investigator — PBRC Co-Principal Investigator; Conrad Earnest, PhD, Study Chair — PBRC Co-Investigator; Catrine Tudor-Locke, PhD, Study Chair — PBRC Co-Investigator; William Johnson, PhD, Study Chair — PBRC Co-Investigator; Jennifer Rood, PhD, Study Chair — PBRC Co-Investigator
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Dorling JL, Hochsmann C, Fearnbach SN, Apolzan JW, Hsia DS, Johannsen NM, Church TS, Martin CK. Initial Weight Change and Long-Term Changes in Weight and Compensation during Supervised Exercise Training. Med Sci Sports Exerc. 2021 Aug 1;53(8):1675-1684. doi: 10.1249/MSS.0000000000002633. PMID 33731664
- [Derived] Martin CK, Johnson WD, Myers CA, Apolzan JW, Earnest CP, Thomas DM, Rood JC, Johannsen NM, Tudor-Locke C, Harris M, Hsia DS, Church TS. Effect of different doses of supervised exercise on food intake, metabolism, and non-exercise physical activity: The E-MECHANIC randomized controlled trial. Am J Clin Nutr. 2019 Sep 1;110(3):583-592. doi: 10.1093/ajcn/nqz054. PMID 31172175
- [Derived] Sarzynski MA, Ruiz-Ramie JJ, Barber JL, Slentz CA, Apolzan JW, McGarrah RW, Harris MN, Church TS, Borja MS, He Y, Oda MN, Martin CK, Kraus WE, Rohatgi A. Effects of Increasing Exercise Intensity and Dose on Multiple Measures of HDL (High-Density Lipoprotein) Function. Arterioscler Thromb Vasc Biol. 2018 Apr;38(4):943-952. doi: 10.1161/ATVBAHA.117.310307. Epub 2018 Feb 8. PMID 29437573
- [Derived] Myers CA, Johnson WD, Earnest CP, Rood JC, Tudor-Locke C, Johannsen NM, Cocreham S, Harris M, Church TS, Martin CK. Examination of mechanisms (E-MECHANIC) of exercise-induced weight compensation: study protocol for a randomized controlled trial. Trials. 2014 Jun 7;15:212. doi: 10.1186/1745-6215-15-212. PMID 24906459

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise Group (20 KKW) | Exercise Group (8 KKW) | Control Group
Started | 67 | 66 | 65
Completed | 51 | 59 | 61
Not Completed | 16 | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Group (20 KKW) | Exercise Group (8 KKW) | Control Group | Total
Number analyzed (Participants) | 51 | 59 | 61 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (12.4) | 48.3 (11.2) | 49.5 (10.8) | 48.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 43 | 45 | 124
  Male | 15 | 16 | 16 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 20 | 21 | 53
  White | 37 | 39 | 38 | 114
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: A Comparison of the Effects of Energy Balance With Three Groups. [Energy Intake, Adjusted DLW]
Description: A comparison of three groups for the effects of energy balance: 1. Healthy Living, 2. Recommended dose exercise, and 3. High dose exercise. Random assignment is determined by chance.
  Healthy Living Group: Information tips on a variety of topics, including stress management, the benefits of eating fruits and vegetables, and other health related matters. This information is sent directly to your cell phone or email address throughout the study. Encouragements are sent to attend monthly seminars on various health topics at Pennington. Maintain a baseline level of exercise throughout the study.
  Recommended Dose Exercise: 3 t0 4 low-intensity sessions per week, each lasting about 30 minutes, at Pennington Fitness and Wellness Center. All exercise will be done on a treadmill.
  High Dose Exercise: 4 to 5 high-intensity session s per week, each lasting about 50-70 minutes, at Pennington Fitness and wellness center. All exercise will be done on the treadmill.
Time Frame: 6 months after screening
Measure: Mean (95% Confidence Interval); unit: kcal/day
Arm/Group | Exercise Group (20 KKW) | Exercise Group (8 KKW) | Control Group
Number analyzed (Participants) | 51 | 59 | 61
kcal/day | 123.6 [64.5 to 182.7] | 90.7 [35.1 to 146.4] | -2.3 [-58.0 to 53.5]

ADVERSE EVENTS:
Arm/Group | Exercise Group (20 KKW) | Exercise Group (8 KKW) | Control Group
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/66 | 0/65
Serious Adverse Events (participants affected / at risk) | 3/67 | 3/66 | 0/65
Other Adverse Events (participants affected / at risk) | 11/67 | 14/66 | 5/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exercise Group (20 KKW) (N=67) | Exercise Group (8 KKW) (N=66) | Control Group (N=65)
pelvis fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
global amnesia (Psychiatric disorders) | 0 | 1 | 0
venous engorgement and orbital swelling (Vascular disorders) | 1 | 0 | 0 — VENOUS ENGORGEMENT AND ORBITAL SWELLING O.D. PRIOR CAROTID ULTRASOUND STUDY AND MRI SUGGEST A-VSHUNT IN RIGHT CAROTID ARTERY SYSTEM
pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0
prostate biopsy positive for malignant cells (Reproductive system and breast disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exercise Group (20 KKW) (N=67) | Exercise Group (8 KKW) (N=66) | Control Group (N=65)
sinus infection/URI (Infections and infestations) | 5 | 6 | 0
basal cell carcinoma removed from ear (Surgical and medical procedures) | 0 | 1 | 0
rotator cuff repair (Surgical and medical procedures) | 0 | 1 | 0 — ARTHROSCOPIC RIGHT SHOULDER ROTATOR CUFF REPAIR
motor vehicle collision (Injury, poisoning and procedural complications) | 0 | 2 | 0 — had brushing to L thigh area
foot pain (Injury, poisoning and procedural complications) | 1 | 1 | 0
pelvic and pudenda pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
laprascopic myomectomy (Surgical and medical procedures) | 0 | 1 | 0
bone fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 — FRACTURED BONE IN LEFT FOOT. OCCURRED WITH MISSTEP ON STAIRS ON CRUISE SHIP.
fell down stairs at work (Injury, poisoning and procedural complications) | 1 | 0 | 0
pain from degenerative disk disease (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
acute chest pain (Cardiac disorders) | 1 | 0 | 0
migraine headaches (Nervous system disorders) | 1 | 0 | 0
light headed and hypotensive (Injury, poisoning and procedural complications) | 1 | 0 | 0
skin abrasions from EKG leads (Injury, poisoning and procedural complications) | 0 | 0 | 1
knee sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 — unrelated to study protocol
ER visit (Gastrointestinal disorders) | 0 | 0 | 1 — COMPLICATIONS WERE FROM REFLUX AND AIRWAY COMPLICATIONS RELIEVED WITH ALBUTERAL AND PROTONIX.
kidney stones (Renal and urinary disorders) | 0 | 0 | 1
intra-abdominal mass found (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No